CLINICAL TRIAL: NCT05112224
Title: Effectiveness of a Health Education Program Using Health Belief Model to Improve Oral Health in School Going Children
Brief Title: A Model-based Health Education Program to Improve Oral Health in School Going Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Responsible Party: Principal Investigator, Mohsen Saffari, Professor, Baqiyatallah Medical Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BMSU.1395.63789
Record Dates: First submitted 2021-10-19; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Oral Health
Keywords: Oral health; Gingival health; Health education; Decayed teeth
MeSH Terms: conditions — Health Education; Dental Caries

STUDY DESIGN:
Intervention Model Description: One group received the intervention and another received the routine program.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The dentist and data analyzer were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Intervention (Experimental): An educational program based on HBM that was conducted using five one-hour sessions.
  Interventions: Behavioral: Education program based on health belief model to improve oral health
- Control (No Intervention): Control group only received the education program provided by the dental clinic.

INTERVENTIONS:
Behavioral: Education program based on health belief model to improve oral health — Five weekly sessions each one lasted for one hour to encourage participants to follow healthy behaviors on oral health.
  Arms: Educational Intervention

SUMMARY:
This was a randomized controlled trial to assess how an education program based on health belief model (HBM) may affect oral health status in the elementary school going children. For this, a convenient sample including 112 school going children aged between 6-12 years old were recruited and randomized into intervention or control groups. Education program consisted five weekly session each lasted for 1 hour approximately. Based on the main constructs of the HBM, each session was organized and a combination of educational methods were used in the intervention group while the control group only received the routine program provided by the dental clinic. Measures such as papillary bleeding index; decayed, missing, filled teeth (DMFT) and a scale based on the HBM were used for data collection. Three months after the intervention the measures were administered again and comparisons between baseline and follow-up were done.

DETAILED DESCRIPTION:
Oral health problems especially dental carries are common in school children and education programs may help to prevent these conditions. The aim of current study was to investigate how an education program based on health belief model (HBM) may improve oral health status of the elementary school children.

One hundred twelve 6-12 year children along with one of their parents assigned into trial and control groups using a randomized controlled trial. For trial group 5 education sessions based on HBM were held, whereas control group only received routine education program delivered by the dental clinic. Decayed, missing, filled teeth (DMFT) score, papillary bleeding index, and HBM questionnaire for oral were used for evaluation of the program. Three month after the intervention reassessment was performed and the changes were measured by student t test as well as analysis of covariance test.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6-12 years old (elementary school going children)
* Attendance of at least one parent (either father or mother) when admission and to take part in the intervention
* Being permanent residents of the enrollment area
* Having medical record in the dental clinic
* Ability to speak and understand Persian

Exclusion Criteria:

* Children with advanced oral diseases or other critical conditions or disabilities
* Those who were using anti-inflammatory agents as a routine
* Those who had used antibiotics in past two weeks
* Children with illiterate parents
* Those on ongoing orthodontic treatments

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Number of Decayed, missing and filled teeth | Five months
  Measured by decayed, missing and filled teeth (DMFT) score
Gingival health | Five months
  Measured by papillary bleeding index
Constructs of health belief model | Five months
  Measured by health belief model (HBM) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen Saffari, PhD., Study Chair — Baqiyatallah Medical Sciences University
Locations (1):
- Baqiyatallah University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No
No sharing.